CLINICAL TRIAL: NCT02060253
Title: A Phase I Clinical Trial of Ganetespib (Heat Shock Protein 90 Inhibitor) in Combination With Paclitaxel, Trastuzumab and Pertuzumab in Human Epidermal Growth Factor Receptor-2 Positive (HER2+) Metastatic Breast Cancer
Brief Title: Ganetespib, Paclitaxel, Trastuzumab and Pertuzumab for Metastatic Human Epidermal Growth Factor Receptor 2 Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Synta Pharmaceuticals Corp. (Industry); New York University Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-168
Record Dates: First submitted 2014-01-30; First posted 2014-02-12 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — STA 9090; Paclitaxel; Taxes; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ganetespib, paclitaxel, and trastuzumab with pertuzumab (Experimental): Patients receive trastuzumab intravenously (IV) over 30 minutes on days 1, 8, 15, and 22, pertuzumab IV over 30 minutes every 3 weeks (only in Part II of the study, starting day 1), paclitaxel IV over 1 hour on days 1, 8, 15, and 22, and ganetespib IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. The MTD for ganetespib in combination with paclitaxel and trastuzumab is 150 mg/m2.
  Interventions: Drug: ganetespib; Drug: paclitaxel; Biological: trastuzumab; Biological: pertuzumab

INTERVENTIONS:
Drug: ganetespib — Given IV
  Other Names: Hsp90 inhibitor STA-9090; STA-9090
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Biological: pertuzumab — Given IV
  Other Names: Perjeta

SUMMARY:
This phase I trial studies the side effects and best dose of ganetespib when given with paclitaxel, trastuzumab and pertuzumab in treating patients with human epidermal growth factor receptor 2 positive (HER2+) metastatic breast cancer (MBC).

DETAILED DESCRIPTION:
This phase I trial studies the side effects and best dose of ganetespib when given with paclitaxel, trastuzumab, pertuzumab in treating patients with human epidermal growth factor receptor 2 positive (HER2+) breast cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or has returned after a period of improvement (metastatic). HER2+ describes cancer cells that have too much of a protein called HER2 on their surface. In normal cells, HER2 helps to control cell growth. When it is made in larger than normal amounts by cancer cells, the cells may grow more quickly and be more likely to spread to other parts of the body.

Ganetespib may stop the growth of tumor cells by blocking some of the proteins needed for cell growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as trastuzumab and pertuzumab, bind to HER2+ cancer cells and may kill them. Giving ganetespib with paclitaxel, trastuzumab, and pertuzumab may be a better treatment for patients with HER2+ breast cancer.

This phase I study has two parts. During the first part of this study, patients with HER2+ MBC receive trastuzumab in combination with ganetespib and paclitaxel to evaluate the safety, toxicity and maximum tolerated dose (MTD) of this triplet regimen. There are dose escalations for ganetespib. Paclitaxel and trastuzumab are administered at standard doses without escalation. Part 1 is ongoing.

During the second part of this study, pertuzumab at standard dose will be added to the triplet regimen of ganetespib, paclitaxel and trastuzumab, using the MTD of ganetespib determined in part one. The MTD of ganetespib and the safety of the four-drug regimen will be evaluated. The MTD for ganetespib in combination with paclitaxel and trastuzumab is 150 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of breast cancer (central confirmation is not required)
* Patients must be at least 18 years of age
* Metastatic or advanced breast cancer that is evaluable OR metastatic or advanced breast cancer that is measurable for response as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of at least 3 months as assessed by the investigator
* Patients with estrogen receptor (ER)+ breast cancer must have received prior treatment with at least one hormone therapy
* Absolute neutrophil count ≥ 1,500 cells/uL
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 9.0g/dL
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Albumin ≥ 3.0 g/dL
* Adequate renal function as defined by a serum creatinine ≤ 1.5 x ULN
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Female subjects of childbearing potential and males must agree to use adequate contraception (e.g., hormonal or barrier method of birth control; abstinence) for the duration of study treatment
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry
* Patients with human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS) are allowed on study if they have an undetectable viral load, cluster of differentiation (CD)4 > 300 and are on a stable highly active antiretroviral therapy (HAART) regimen for 1 month prior to study enrollment
* Patients are required to have HER2+ breast cancer defined as a fluorescent in situ hybridization (FISH)- ratio of >= 2.0 or immunohistochemistry (IHC) 3+
* Patients for the triplet regimen (ganetespib, paclitaxel, trastuzumab):

  * Any number of prior chemotherapies or biological therapies are allowed, patients are required to have prior treatment with pertuzumab and ado-trastuzumab emtansine with the exceptions listed below:

    * Metastatic patients who have not received prior pertuzumab are eligible if: heavily pretreated prior to Food and Drug Administration (FDA) approval of pertuzumab (08-Jun-2012) for first line treatment of HER2+ MBC
    * Metastatic patients who have not received ado-trastuzumab emtansine are eligible if: heavily pretreated prior to FDA approval of ado-trastuzumab emtansine (22-Feb-2013) for the treatment of patients with HER2+ MBC who previously received trastuzumab and a taxane, separately or in combination
* Patients for the triplet regimen + pertuzumab:

  * Prior hormonal therapy for ER+ and/or PR+ HER2+ disease in the metastatic setting is allowed.
  * Prior T-DM1 in the metastatic setting is allowed if patients have progressed within 6 months after treatment for early-stage disease.
* No prior history of intolerance or hypersensitivity to trastuzumab and/or adverse events related to trastuzumab, murine proteins, or any of the excipients that resulted in trastuzumab being permanently discontinued

Exclusion Criteria:

* Fewer than 21 days since last anti-tumor therapy, including chemotherapy, biologic except trastuzumab, experimental, immune, radiotherapy for the treatment of breast cancer, with the following exceptions:

  * Hormone therapy
  * Palliative radiation therapy involving =< 25% of marrow-bearing bone is allowed if completed within >= 14 days prior to first study treatment
* Surgery, radiotherapy, or lesion ablative procedure to the only area of measurable/evaluable disease
* Major surgery within 4 weeks prior to first dose of ganetespib
* Poor venous access for study drug administration

  * Study drug administration via indwelling catheters is allowed only if the catheter is made of silicone material
* No prior chemotherapy in the metastatic setting is allowed.
* Prior pertuzumab is not allowed in the metastatic setting. Pertuzumab given in the neoadjuvant and/or adjuvant setting is allowed.
* History of intolerance or hypersensitivity to trastuzumab and/or pertuzumab
* Adverse events related to trastuzumab, murine proteins, or any of the excipients that resulted in trastuzumab being permanently discontinued
* History of severe (grade 3 or 4) allergic or hypersensitivity reactions to excipients (e.g., polyethylene glycol [PEG] 300 and polysorbate 80)
* History of intolerance or hypersensitivity to paclitaxel and/or adverse events related to paclitaxel that resulted in paclitaxel being permanently discontinued
* Peripheral neuropathy of grade >= 2 per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, at the time of or within 3 weeks prior to the first study therapy
* Baseline QTc > 470 msec (average of triplicate ECG recordings); a consistent method of QTc calculation must be used for each patient's QTc measurements. QTcF (Fridericia's formula) is preferred
* Use of medications that have been linked to the occurrence of torsades de pointes

  * Patients will be eligible for the study if they discontinue any of the listed medications two weeks prior to registration and study enrollment
  * Stable regimen of antidepressants of the SSRI class is allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline and fluoxetine)
* Left ventricular ejection fraction (EF) < 50% at baseline
* Serum potassium, magnesium, and calcium levels (corrected for albumin) outside the laboratory's reference range despite correction
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation)
* Women who are pregnant or lactating
* Current known active infection with HIV, hepatitis B or C viruses
* Uncontrolled systemic disease (e.g., clinically significant cardiac, pulmonary or metabolic disease)
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results in the judgment of the investigator
* History of clinically significant cardiac dysfunction, including:

  * Unstable angina
  * Unstable atrial fibrillation
  * Symptomatic bradycardia
  * Indwelling temporary pacemaker
  * History of MI within 6 months prior to first study treatment
  * History of symptomatic CHF (grade > 3 by NCI CTCAE or Class > II by New York Heart Association (NYHA) criteria
  * Ventricular tachycardia or a supraventricular tachycardia that requires treatment with a Class 1a antiarrhythmic drug (eg quinidine, procainamide, disopyramide) or Class III antiarrhythmic drug (eg sotalol, amiodarone, dofetilide). Use of other antiarrhythmic drugs is permitted
  * Second or third degree atrioventricular (AV) block unless treated with a permanent pacemaker
  * Complete left bundle branch block (LBBB)
  * History of long QT syndrome or a family member with this condition
* Brain metastases that are:

  * Progressive or
  * Have required any type of therapy (including radiation, surgery or steroids) to control symptoms from brain metastases within 60 days prior to the first study treatment
* History of an invasive second primary malignancy diagnosed within the previous 3 years, except for appropriately treated stage I endometrial or cervical carcinoma or prostate carcinoma treated surgically, and non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended Phase II dose of ganetespib plus paclitaxel plus trastuzumab and pertuzumab | 28 days

SECONDARY OUTCOMES:
Objective Response Rate | Up to 2 years
  Defined as the percentage of patients who have achieved complete response or partial response assessed based on Response evaluation criteria in solid tumors 1.1 (RECIST 1.1).
Clinical benefit rate | Up to 2 years
  Defined as the percentage of patients who have achieved complete response, partial response, or stable disease for at least 24 weeks assessed based on RECIST 1.1.
Duration of response | Up to 2 years
  The duration of response is measured from the time of response to disease progression.
Progression-free survival (PFS) | Up to 2 years
  The median time of progression-free survival will be calculated.

OTHER OUTCOMES:
PK parameters of paclitaxel (such as area under the curve and maximum concentration) | Pre-dose, 0.5, 1, 1.5, 2, 4, 7, 21, 24, 27, and 31 hours
  Will be examined descriptively to evaluate the effect of ganetespib on the paclitaxel absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Shanu Modi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - NYU Cancer Institute, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Jhaveri K, Wang R, Teplinsky E, Chandarlapaty S, Solit D, Cadoo K, Speyer J, D'Andrea G, Adams S, Patil S, Haque S, O'Neill T, Friedman K, Esteva FJ, Hudis C, Modi S. A phase I trial of ganetespib in combination with paclitaxel and trastuzumab in patients with human epidermal growth factor receptor-2 (HER2)-positive metastatic breast cancer. Breast Cancer Res. 2017 Aug 2;19(1):89. doi: 10.1186/s13058-017-0879-5. PMID 28764748
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/